CLINICAL TRIAL: NCT03041207
Title: Decreasing Antibiotic Use in Infants With Suspected Ventilator-associated Infection
Acronym: VAIN2
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: HM20009140
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Ventilator Associated Pneumonia; Nosocomial Infections in Children; Microbial Colonization
Keywords: ventilator associated infection; ventilator associated pneumonia; ventilator associated tracheitis; Lower respiratory infection
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Communicable Diseases | interventions — Growth and Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-antibiotic guideline: Infants for whom antibiotics have been initiated for suspected ventilator-associated infection prior to the implementation of the antibiotic guideline
  Interventions: Behavioral: Development and implementation of an antibiotic guideline
- After antibiotic guideline implementation: Infants for whom antibiotics have been initiated for suspected ventilator-associated infection after the implementation of the antibiotic guideline
  Interventions: Behavioral: Development and implementation of an antibiotic guideline
- Microbiome Study Group: Infants intubated and anticipated to require mechanical ventilation for at least several days

INTERVENTIONS:
Behavioral: Development and implementation of an antibiotic guideline — A consensus conference will develop and then implement a guideline for stopping vs. continuing antibiotics in infants with suspected ventilator-associated infection
  Groups: After antibiotic guideline implementation; Pre-antibiotic guideline

SUMMARY:
This is a prospective study with three specific aims: (1) To convene a consensus conference to develop a guideline for antibiotic use in infants (age < 3 yrs) with suspected ventilator-associated infection; (2) To evaluate outcomes before and after implementation of the antibiotic guideline; (3) To evaluate changes in the tracheal microbiome over the course of mechanical ventilation

DETAILED DESCRIPTION:
In 2011 the Centers for Disease Control (CDC) estimated antibiotic-resistant infections resulted in $20 billion in excess healthcare costs and more than 100,000 unnecessary deaths in the U.S. alone. Ventilator-associated infections (VAI) are the most commonly diagnosed hospital-acquired infections in the pediatric intensive care unit (PICU) and account for more than half of all antibiotic use. We believe the diagnosis is often in error and that much of the antibiotic use is unnecessary. Initiating broad-spectrum antibiotics is routine when VAI or other infection is suspected in the child on mechanical ventilation, but our data show when all other cultures are negative at 48-72 hours antibiotics are frequently still continued based on identification of bacteria in respiratory secretion cultures. The investigators have previously shown, however, that identification of bacteria in respiratory secretion cultures is common in asymptomatic children and continuing antibiotics on the basis of a "positive" respiratory secretion culture is not associated with a shorter hospital stay or improved survival.

Antibiotics are not benign. Antibiotics are expensive, have disproportionate adverse effects in younger children, often require placement of catheters that are themselves potential sources of infection, and their overuse has been associated with increasing resistance worldwide. Antibiotic exposure in young children has been associated with increased risk for obesity, types 1 and 2 diabetes, inflammatory bowel diseases, celiac disease, allergies, and asthma. Mouse studies have found that early antibiotic exposure disrupts the development of the early-life gut bacterial composition (microbiome), leading to metabolic perturbations that affect fat deposition and may alter normal immunologic development.

There is no diagnostic test for VAI and distinguishing tracheal bacterial colonization from actual infection is not straightforward. The normal lung is essentially sterile but placement of an endotracheal tube (ETT) compromises the lung's ability to clear aspirated secretions and allows a direct route for bacterial contamination from the mouth and throat. The resultant tracheal bacterial composition (the "microbiome") is largely unstudied but preliminary research suggests it consists of small numbers of a wide diversity of bacteria originating from the mouth. Loss of this bacterial diversity in conjunction with proliferation of pathological bacteria is thought to herald the conversion from colonization to infection.

The investigators believe that a positive respiratory culture alone in the absence of other indicators of infection is insufficient justification for continuing antibiotics and, consequently, much of the antibiotic use in VAI is both unnecessary and potentially harmful. To critically evaluate this belief and potentially decrease the use of unnecessary antibiotics we propose the following:

Aim 1: To develop a guideline to assess the likelihood of VAI and discontinue antibiotics when the risk is judged to be low Hypothesis 1.1: Using an iterative process PICU doctors can reach consensus on criteria to assess the likelihood of VAI and discontinue antibiotics when the risk of VAI is judged to be low

Aim 2: To assess the efficacy and safety of discontinuing antibiotics in children judged to have a low risk of VAI Hypothesis 2.1: Discontinuing antibiotics at 48-72 hours in children judged to have a low risk of VAI will result in fewer total days on antibiotics with no difference in survival, numbers of subsequent infection episodes, duration of need for mechanical ventilation and length of stay in the PICU compared to care prior to the implementation of the guideline.

Aim 3: To describe the longitudinal changes in the tracheal bacterial composition (the "microbiome") in children on mechanical ventilation Hypothesis 3.1: Loss of diversity in the tracheal microbiome will predate clinical signs and symptoms of VAI.

Hypothesis 3.2: Emergence of a dominant bacterial pathogen in the tracheal microbiome will be associated with clinical signs and symptoms of VAI.

Decreasing unnecessary antibiotic use has important implications for public health. Pediatric intensive care medicine is running out of effective antibiotics while also exposing our children to antibiotic risks, many of which are only now beginning to be understood. Avoidance of unnecessary antibiotic exposure in young children is critical and would be facilitated by a rational guideline for assessment of the risk and appropriate treatment for suspected VAI. As VAI is the most common reason for antibiotic use in the PICU, it is an obvious target for more careful antibiotic stewardship. Better understanding of the normal tracheal microbiome after placement of an endotracheal tube would also inform future decisions regarding appropriate antibiotic use when VAI is suspected. The most effective means of decreasing antibiotic resistance is avoidance of unnecessary use.

ELIGIBILITY:
Inclusion Criteria:

* Age newborn -- 3 years in the Pediatric ICU
* on invasive mechanical ventilation > 48 hours
* evaluation for ventilator-associated infection that includes respiratory secretion cultures and microscopic evaluation of the gram-stained specimen
* antibiotics initiated for suspected ventilator-associated or other infection

Exclusion Criteria:

* Immune compromise --Other positive cultures (blood, urine, etc.) for which antibiotic continuation is appropriate

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants 0 - 3 years of age who have undergone a tracheal aspirate culture for suspected ventilator-associated infection and have had antibiotics initiated at that time.
Sampling Method: Non-Probability Sample
Enrollment: 555 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Pediatric ICU-free days at 28 days | 28 days after study enrollment
  28 - number of days in PICU (death = 0 free days)

SECONDARY OUTCOMES:
Antibiotic days in PICU | 28 days after study enrollment
  total number of antibiotic days with each antibiotic on each day = 1 antibiotic day (e.g., 3 antibiotics in one day = 3 antibiotic days)
Ventilator-free days at 28 days | 28 days after study enrollment
  28 - days on mechanical ventilation in PICU (death = 0 free days)
Infection and sepsis episodes | 28 days after study enrollment
  The number of infection and/or sepsis episodes after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Douglas F Willson, MD, Principal Investigator — Virginia Commonwealth University
Locations (23):
- United States (22):
  - Banner University Medical Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Miami Health System - Holtz Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta - Egleston Hospital, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - St. Louis Children's Hospital - Washington University, St Louis, Missouri
  - Children's Hospital of Buffalo, Buffalo, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No